CLINICAL TRIAL: NCT04291092
Title: Camrelizumab Combined With Chemotherapy and Local Treatment in Non-small Cell Lung Cancer Patients With Brain Metastasis, a Single-arm, Multi-center, Open-labeled Phase II Clinical Trial
Brief Title: Camrelizumab Combined With Local Treatment in NSCLC Patients With BM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, GongLei, Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYJ20200101-1
Record Dates: First submitted 2020-01-08; First posted 2020-03-02 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: NSCLC Stage IV; Brain Metastases; Immunotherapy
Keywords: lung cancer; Brain Metastases; Camrelizumab; WBRT; SRS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — Immunotherapy; camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental): single-arm
  Interventions: Drug: Immunotherapy; Radiation: WBRT; Drug: Chemotherapy

INTERVENTIONS:
Drug: Immunotherapy — Immunotherapy for brain metastasis
  Other Names: Camrelizumab
Radiation: WBRT — local therapy for brain metastasis
  Other Names: SRS
Drug: Chemotherapy — Chemotherapy for brain metastasis

SUMMARY:
To evaluate the efficacy and safety of Camrelizumab Combined with Chemotherapy and Local Treatment in non-small cell lung cancer with brain metastases.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Camrelizumab Combined with Chemotherapy and Local Treatment of brain metastases (WBRT, r-knife, SRS, etc.) in non-small cell lung cancer patients with brain metastases .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. ECOG is 0-1;
3. Non-small cell lung cancer confirmed by histology; EGFR、ALK and ROS1 negative;
4. The presence of brain metastases as determined by imaging, with unlimited numbers, the intracranial lesions had a maximum diameter of ≥ 0.5cm，allowing the presence of clinical symptoms of brain metastases;
5. According to RECIST 1.1, there is at least one measurable extracranial and intracranial target lesion each;
6. Sign informed consent and agree to collect the clinical efficacy and information of the patient.

Exclusion Criteria:

1. Immunotherapeutic contraindications (including long-term use of hormones, history of radiation pneumonia, etc.)
2. Active autoimmune diseases (e.g. vitiligo, psoriasis, hypothyroidism requiring hormone replacement therapy, etc.)
3. Patients with active hepatitis B or C, HIV, active tuberculosis, etc.;
4. Active infections requiring antimicrobial therapy (e.g. antimicrobial, antiviral, antifungal);
5. History of known allogeneic organ transplantation and history of in vivo hematopoietic stem cell transplantation;
6. Patients with interstitial lung disease or previous history of interstitial pneumonia;
7. Having a history of substance abuse and unable to abstain from it or having mental disorders;
8. who have participated in other clinical trials of antitumor drugs within 4 weeks before entering the group;
9. Having used PD-1/PD-L1 and other immunotherapy drugs before entering the group;
10. previous or concurrent with other untreated malignancies, except for cured basal cell carcinoma of the skin, carcinoma of the cervix in situ and superficial bladder cancer;
11. (a) Pregnant or lactating women; those with fertility who are unwilling or unable to take effective contraception;
12. The researchers judged other situations that might affect the conduct of clinical studies and the determination of their findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
6 month progression-free survival rate | 6 month
  6 month progression-free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xu Y, Chen K, Xu Y, Li H, Huang Z, Lu H, Huang D, Yu S, Han N, Gong L, Qin J, Chen J, Xie F, Hong W, Lin X, Cheng F, Luo X, Fan Y. Brain radiotherapy combined with camrelizumab and platinum-doublet chemotherapy for previously untreated advanced non-small-cell lung cancer with brain metastases (C-Brain): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2025 Jan;26(1):74-84. doi: 10.1016/S1470-2045(24)00643-0. PMID 39756446